CLINICAL TRIAL: NCT05013138
Title: Addressing ACEs Among Hispanic Caregivers in a Pediatric Primary Care Population to Improve Child Health and Decrease Early Adversity
Brief Title: Caregiver Adverse Childhood Experiences (ACEs) in Pediatric Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Abigail Lott, Assistant Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002897; 1R49CE003072-01-4 (Other Grant/Funding Number: CDC); 1R49CE003072-01 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Child Development
Keywords: Adverse Childhood Experiences
MeSH Terms: interventions — N-(2-acetamido)-2-aminoethanesulfonic acid

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial. Randomization occurs at the provider level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (Active Comparator): During the study period, standard of care providers will continue to provide standard of care treatment(s); however, families receiving care from the standard of care providers will complete all study surveys. Instead of ACEs training, standard of care providers will undergo training on study procedures including obtaining survey instruments from caregivers and proper storage of survey instruments. This training will stress the importance of not reviewing caregiver ACE scores and minimizing possible treatment contamination. However, standard of care providers will still be able to provide resources to the families as part of standard of care.
  Interventions: Behavioral: Training on study procedures
- Intervention Arm (Experimental): Intervention providers will undergo training for ACEs screening and discussion. Eligible families will be enrolled into the study at the intake of their child's 4-month, 6-month, 9-month, 15-month, or 18-month well child check. Caregivers will complete the intake surveys including demographics, caregiver ACEs, resilience, warmth, PTSD, and depression. The providers will lead a discussion regarding the impact of caregiver ACEs. Patients will be contacted 1-week, 6-months, and 18-months following their enrollment to obtain repeat measures of the survey instruments. At the 18-month time point, the electronic medical record (EMR) will be queried to obtain outcome measures.
  Interventions: Behavioral: Training for ACEs and study procedures

INTERVENTIONS:
Behavioral: Training for ACEs and study procedures — The providers will lead a resilience-based conversation discussion regarding the impact of caregiver ACEs, after receiving training for ACEs and study procedures.
  The first training component will provide an overview of ACEs using the ACE Interface Training. The second training component will address the implementation of the caregiver ACEs screening in the clinic.
  Arms: Intervention Arm
Behavioral: Training on study procedures — Instead of ACEs training, standard of care providers will undergo training on study procedures including obtaining survey instruments from caregivers and proper storage of survey instruments. This training will stress the importance of not reviewing caregiver ACE scores and minimizing possible treatment contamination.
  Arms: Standard of Care Arm

SUMMARY:
This longitudinal study will evaluate if increased caregiver awareness of their own ACEs through provider-led discussions will lead to improved child health via fewer emergency department, urgent care visits and missed primary care appointments.

DETAILED DESCRIPTION:
This longitudinal study will examine whether screening for caregiver adverse childhood experiences (ACEs) and a provider-led discussion of how exposure to ACEs impacts parenting will improve child health outcomes over an 18 month period compared to treatment as usual in a pediatric primary care setting during infant well-child visits. Child health outcomes examined will be rates of emergency department and urgent care visits. Potential protective factors, including parental warmth and resilience will also be examined. The population being studied will include caregivers to infants (ranging 1 week-18 months) receiving care at Mercy Care Clinic (MCC) in Chamblee, Georgia (GA), which primarily serves Hispanic families. Contact will be made by approaching patients present for an infant well-child visit in the clinic. Informed consent will be obtained by a study staff member in the waiting room of the Mercy Care Chamblee Clinic. Electronic or written consent (in English or Spanish based on patient preference) will be obtained. This is not a no-contact study. Data will not be publicly available, but deidentified data will be available upon request beginning 12 months after the study is completed. Only direct study staff will have access to identifying information for participants. Privacy of existing data is not a concern. Interactions will include participant's filling out surveys (or having surveys read aloud to them in their preferred language) and chart review. Those participants who meet with providers randomized to the ACEs discussion will also have a short discussion with their provider about any experienced ACEs and forms of resilience they note on the surveys. Data will be collected in the clinic setting and for follow-up visits by phone or internet based on participant preference.

Topics assessed will include exposure to adverse experiences in childhood, depression and posttraumatic stress disorder symptoms, resilience, and parenting. Each assessment will take less than one hour to complete. All participants will be given a subject identification (ID) number upon consent and all data will be deidentified and only associated with that ID number for the remainder of the study. Medical records will be examined for appointment confirmation (eligibility) and for infant medical visits over the course of the study (outcome variable) and only study staff will have access to identifiable information.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers will be eligible to enroll in the study if they bring children to the MCC for either a 4-month, 6-month, 9-month, 15-month, or 18-month WCC. Notably, we anticipate the majority of participants to be of Hispanic origin and many to be exclusively Spanish-speaking. All Research Assistants (RAs) working directly with caregivers will be bilingual according to Emory Spanish fluency testing. We will solicit expert opinion from faculty that work with these communities and the staff of MCC that work with these patients on a regular basis.

Exclusion Criteria:

* Caregivers will be excluded if they are unable to speak and read either English or Spanish. Caregivers will also be excluded if they have already been enrolled in the study protocol via another child or prior WCC. Caregivers who are under the age of 18 years will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Number of emergency department (ED) visits documented in chart at 18 months post-intervention | 18 months post-intervention
  Number of emergency department (ED) visits documented in chart from baseline to 18 months post-intervention
Number or urgent care (UC) visits documented in chart at 18 months post-intervention | 18 months post-intervention
  Number or urgent care (UC) visits documented in chart from baseline to18 months post-intervention
Number of medical visits at Mercy Care at 18 months post-intervention | 18 months post-intervention
  Number of medical visits at Mercy Care over the course of the study period will be obtained from baseline to 18 months post-intervention.

SECONDARY OUTCOMES:
Change in Primary Care PTSD score for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) from Baseline Caregiver's PTSD symptoms due to ACEs screening | Baseline, 1 week post-intervention, 6 months follow up, 18 months follow up
  The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) is a 5-item screen designed for use in primary care will assess for presence of PTSD symptoms. This measure will be used to evaluate baseline PTSD symptoms and changes in symptoms as a result of ACEs intervention. The total score is the sum of "yes" responses. Possible range is 0 to 5. Lower score correlates with better outcome.
Change in Brief Resilience Scale score from baseline | Baseline, 6 months follow up, 18 months follow up
  The investigators will utilize the Brief Resilience Scale (BRS) that focuses on an individual's ability to bounce back from stress. It includes 6 items for caregivers to answer, with the total ranging from 6-30. Higher scores indicate greater levels of resilience. The Brief Resilience Score will be examined as a potential mediator between provider-led ACEs discussion and child health outcomes.
Change in Parenting Questionnaire (PQ) warmth subscale (PQ-warmth) score from Baseline | Baseline, 6 months follow up, 18 months follow up
  The PQ (McCabe & Clark, 1999 )is a 50-item parent self-report of parenting practices, including warmth; that was modified to include only 13 items relevant for young children. The warmth subscale total ranges from 13-65. Higher scores indicate greater parental warmth. Parental warmth will be examined as a potential mediator between provider-led ACEs discussion and child health outcomes.
Rate of referrals to Division of Family and Child Services (DFACS) at 18 months post-intervention | 18 months post-intervention
  Number of referrals to DFACS will be obtained during follow up period (from baseline to 18 months post-intervention).
Attendance at well child check (WCC) visits at 18 months post-intervention | 18 months post-intervention
  Number of visits at WCC be obtained during follow up period (from baseline to 18 months post-intervention).
Rate of referrals to non-DFACS services at 18 months post-intervention | 18 months post-intervention
  Number of referrals to non-DFACS will be obtained during follow up period (from baseline to 18 months post-intervention).
Rate of clinic-based social worker visits at 18 months post-intervention | 18 months post-intervention
  Number of clinic-based social worker visits will be obtained during follow up period (from baseline to 18 months post-intervention).
Subjective experience of caregiver ACEs screening on clinic staff at baseline | Baseline
  It will be assessed with a brief qualitative questionnaire. The investigators will ask if staff felt that the ACEs screening negatively/neutral/positively impacted patient experience and staff experience of well-child visits. Scores will range from -1 to +1 for each item and total scores may range from -2 to +2 with higher scores reflecting a more positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Lott, PhD, ABPP, Principal Investigator — Emory University
Locations (1):
- Mercy Care Chamblee, Chamblee, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will not be publicly available, but deidentified data will be available upon request beginning 12 months after the study is completed. Deidentified data files, the data dictionary, and the final protocol will be shared via Emory Dataverse, which is a long-term repository hosted within the University of North Carolina (UNC) Dataverse (listed in the global Registry of Research Data Repositories [re3data.org]).
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 12 months after this study is complete.
Access Criteria: Data will be available for sharing with investigators who email the PI to request access to the deidentified data for any type of analysis.

DOCUMENTS (1):
  • Informed Consent Form (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05013138/ICF_000.pdf